CLINICAL TRIAL: NCT04283357
Title: Effect of Virtual Reality on Pes Planus
Brief Title: Comparison Of Effects Virtual Reality and Short Foot Exercises On Balance and Performance in Pes Planus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Tezel Yıldırım Şahan, Director, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019.06.10
Record Dates: First submitted 2019-07-05; First posted 2020-02-25 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Virtual Reality
Keywords: virtual reality; foot posture; navicular drop; short foot exercise
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: One group only are treated with short foot exercises. Second group are treated with short foot exercises and virtual reality.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Active Comparator): One group only treated with short foot exercises.
  Interventions: Other: Exercise
- Virtual Reality Group (Active Comparator): The second group treated with virtual reality
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Other: Exercise — Short Foot Exercises
  Arms: Exercise Group
Device: Virtual Reality — Exercise with virtual reality
  Arms: Virtual Reality Group

SUMMARY:
Virtual reality exercises have become increasingly popular in recent years. After the increase in usage areas in daily life, its use in healthcare has become widespread. Flatfoot is one of the orthopedic problems with high prevalence, especially in young individuals. In the literature, conservative treatment methods of flat soles are mentioned as exercise, shoe modifications, and orthotic methods. In the study, it is planned to investigate whether individuals with flat-footed virtual reality exercises contribute to conservative treatment.

The aim of this study was to investigate the effect of virtual reality exercises on individuals with pes planus.

DETAILED DESCRIPTION:
To show whether virtual reality exercises will contribute to decrease of flat footing, improvement of balance and increase of performance of individuals with flat foot.

ELIGIBILITY:
Inclusion Criteria:

* Have pes planus,
* Volunteer for this study,
* Climb 10 stairs independently,
* Can stand one single leg

Exclusion Criteria:

* History of trauma, fracture or operation of the foot, knee, and hip that will affect the foot
* Having visual, hearing and mental problems that prevent participation in virtual reality exercises,
* Being diagnosed with orthopedic or neurological problems that prevent standing on a single leg

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
comparison of exercise and virtual reality treatment on balance | 15 minute
  Y balance test measure with second (sn)

SECONDARY OUTCOMES:
Effect of exercise on performance | 10 minute
  10 step test measure with minute
Navicular Drop Test | 5 minute
  Measure of navicular tubercul from floor measure with santimeter(cm)
Femoral anteversion test | 5 minute
  measure of hip internal rotation movement actively measure with universal goniometer (degree)

CONTACTS AND LOCATIONS:
Overall Officials: Cevher Demirci, Dr, Study Director — Kırıkkale University
Locations (1):
- Kırıkkale University, Kırıkkale, Yahşihan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The subjects were randomly assigned to one of the groups using an online random allocation software program. All groups were taken into a 4-week treatment program. At the end of the treatment process, it was given to subjects including VR and SF program aiming foot muscles.

REFERENCES:
- [Derived] Yildirim Sahan T, Aydogan Arslan S, Demirci C, Oktas B, Sertel M. Comparison Of Short-Term Effects Of Virtual Reality and Short Foot Exercises In Pes Planus. Foot (Edinb). 2021 Jun;47:101778. doi: 10.1016/j.foot.2021.101778. Epub 2021 Jan 21. PMID 33962115
- See also: Spring ligament complex and posterior tibial tendon: MR anatomy and findings in acquired adult flatfoot deformity — http://www.thieme-connect.com/products/ejournals/abstract/10.1055/s-0036-1580616
- See also: Differences in Static- and Dynamic-Balance Task Performance After 4 Weeks of Intrinsic-Foot-Muscle Training: The Short-Foot Exercise Versus the Towel-Curl Exercise — http://journals.humankinetics.com/view/journals/jsr/21/4/article-p327.xml
- See also: Quality of Life in Adult Population with Flat Feet — http://www.ijhsr.org/IJHSR_Vol.10_Issue.2_Feb2020/IJHSR_Abstract.030.html